CLINICAL TRIAL: NCT01239277
Title: Combined Nutrient Intake and Muscle Protein Synthesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MEC 10-3-080
Record Dates: First submitted 2010-11-10; First posted 2010-11-11 (Estimated); Last update posted 2011-09-14 (Estimated); Status verified 2011-09

CONDITIONS: Aging
Keywords: muscle; FSR; protein; carbohydrate; leucine
MeSH Terms: interventions — Proteins; Carbohydrates; Leucine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- protein (elderly) (Experimental)
  Interventions: Other: protein
- protein and carbohydrate (elderly) (Experimental)
  Interventions: Other: protein and carbohydrate
- protein and carbohydrate (young) (Experimental)
  Interventions: Other: protein and carbohydrate
- protein and leucine (elderly) (Experimental)
  Interventions: Other: protein and leucine

INTERVENTIONS:
Other: protein — 20g protein
  Arms: protein (elderly)
Other: protein and carbohydrate — 20g protein and 20g carbohydrate
  Arms: protein and carbohydrate (elderly); protein and carbohydrate (young)
Other: protein and leucine — 20g protein, 2.5g leucine
  Arms: protein and leucine (elderly)

SUMMARY:
Dietary intervention to prevent sarcopenia in elderly people. The objective of this study is to test whether combined nutrient intake plays an important role in stimulation of the muscle protein growth in elderly people; and whether it represent effective strategies to overcome the impaired muscle protein synthesis in elderly when compared with young subjects.

ELIGIBILITY:
Inclusion Criteria:

* males
* 70-85 years or 18-30 years
* BMI < 30

Exclusion Criteria:

* Type II diabetes
* All co morbidities interacting with mobility and muscle metabolism of the lower limbs
* Use of anticoagulants
* Patients suffering from Phenylketonuria
* Participation in any regular exercise programme

Ages: 70 Years to 85 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 48 (Actual)
Dates: Start 2011-01; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Muscle protein synthesis | 6 h postprandial period
  Muscle protein synthesis will be expressed as fractional synthetic rate (FSR) by dividing the increment in enrichment in the product, i.e. protein-bound C13phe, by the enrichment of the precursor (=plasma availability).

CONTACTS AND LOCATIONS:
Overall Officials: A. de Lange, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Universiteit Maastricht, Bewegingswetenschappen, Maastricht, Limburg, Netherlands

REFERENCES:
- See also: Information about research performed by the Maastricht Muscle Metabolism group at MUMC — http://www.m3-research.nl